CLINICAL TRIAL: NCT05763173
Title: The Diagnostic Value of Lung Ultrashort Echo Time MRI for Potential Lung Metastases in Children With Hepatoblastoma
Brief Title: Evaluation of Lung Metastases Based on Ultrashort Echo Time MRI
Status: Completed | Type: Observational
Sponsor: RenJi Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: LY2022-064-B
Record Dates: First submitted 2023-02-28; First posted 2023-03-10 (Actual); Last update posted 2024-04-18 (Actual); Status verified 2024-04

CONDITIONS: Hepatoblastoma; Radiology
MeSH Terms: conditions — Hepatoblastoma

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Months
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Analyze the diagnostic efficiency (including performance, diameter, and location of nodules) of UTE-MRI in lung metastases of hepatoblastoma with chest CT as gold standard

ELIGIBILITY:
Inclusion Criteria:

* Children diagnosed as hepatoblastoma (including treated with neoadjuvant chemotherapy but not surgery)
* Recent chest CT scan (within 14 days)
* No MRI contraindications
* The guardian of the children are willing to undergo the examination after full communication and informed consent

Exclusion Criteria:

* MRI contraindications (including but not limited to: contrast medium allergy; Claustrophobia;Metal implants;chronic kidney disease≥stage 3 (glomerular filtration rate < 60 mL min-1 (1.73 m2)-1))
* Patients with hepatoblastoma aged 14 years and above
* Children after surgery for hepatoblastoma
* Application of any contrast medium within 24 h before the MRI and/or CT examinations
* There is a concomitant medical condition (e.g. poorly controlled hypertension, severe diabetes, neurological or psychiatric illness, etc.) or any other condition that would seriously endangers the subject's safety, may confuse the study results, or may interfere with the subject's completion of the study according to the investigator's judgment.

Max Age: 14 Years | Sex: All
Age Groups: Child
Study Population: Children diagnosed as hepatoblastoma
Sampling Method: Non-Probability Sample
Enrollment: 65 (Actual)
Dates: Start 2023-01-01 (Actual); Primary Completion 2024-02-29 (Actual); Study Completion 2024-02-29 (Actual)

PRIMARY OUTCOMES:
UTE-MRI assessment of lung metastases with chest CT as gold standard | Baseline to 14 days
  Analyze the diagnostic efficiency (including performance, diameter, and location of nodules) of UTE-MRI in lung metastases of hepatoblastoma.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Radiology, Renji Hospital, School of Medicine, Shanghai Jiaotong University, Shanghai, Shanghai Municipality, China